CLINICAL TRIAL: NCT04275609
Title: The Efficiency of Writing Endoscopic Reports by Artificial Intelligence and Physicians: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2020SDU-QILU-G002
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Gastrointestinal Disease
Keywords: Endoscopic Report; Artificial Intelligence; Gastrointestinal Disease; Writing Efficiency
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Intelligence generating endoscopic report (Experimental): In this group, the endoscopic report was generated by artificial intelligence (AI) based on the structured diagnostic report generation system.
  Interventions: Other: AI generated report
- Physicians writing endoscopic report (Active Comparator): In this group, the endoscopic report was writing by physicians.
  Interventions: Other: physicians writing report

INTERVENTIONS:
Other: AI generated report — After the endoscopic procedure, the physicians click the structured reporting button of computer to automatically complete the report through the structured diagnostic report generation system. The physicians only make minor corrections to the report.
  Arms: Artificial Intelligence generating endoscopic report
Other: physicians writing report — After the endoscopic procedure, the physicians writing the report in computer according the procedure.
  Arms: Physicians writing endoscopic report

SUMMARY:
The purpose of this study is to compare the efficiency of writing endoscopic reports by artificial intelligence and physicians through a randomized controlled trial.

DETAILED DESCRIPTION:
Digestive endoscopy permits early detection of gastrointestinal diseases and improving the patients' quality of life. However, writing endoscopic report takes a lot of manpower and time, reducing the efficiency of endoscopy. Our center has developed a structured diagnostic report generation system for digestive endoscopy, which can generates the report by artificial intelligence. Here, we compare the efficiency of writing endoscopic reports by artificial intelligence and physicians through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 80 years；
* patients undergoing gastroscopy and colonoscopy examination with anesthesia；
* patients able to give informed consent

Exclusion Criteria:

* patients with the contraindications to endoscopic examination;
* a history of gastrointestinal cancers;
* allergic to anaesthetics in previous medical history;
* the endoscopic procedure cannot be completed due to stenosis, obstruction, solid food or complications of anaesthesia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-20 (Estimated); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
The time spent writing reports | Intraoperative
  Sum of the time for writing gastroscopic report and colonoscopic report。

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University